CLINICAL TRIAL: NCT03783702
Title: Multi-institutional, Randomized Controlled Trial Assessing Opioid Use and Analgesic Requirements After Endoscopic Sinus Surgery
Brief Title: Pain Control Following Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Mayo Clinic (Other); Vanderbilt University Medical Center (Other); Albert Einstein College of Medicine (Other); University of British Columbia (Other); Endeavor Health (Other)
Responsible Party: Principal Investigator, Peter Hwang, Principal Investigator, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46384
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Sinusitis; Opioid Use; Opioid Abuse; Narcotic Use; Otolaryngologic Disease; Postoperative Pain; Pain
MeSH Terms: conditions — Sinusitis; Opioid-Related Disorders; Otorhinolaryngologic Diseases; Pain, Postoperative; Pain | interventions — Oxycodone; Magnesium; Tablets; Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two groups: one will receive acetaminophen and oxycodone while the other will receive acetaminophen, ibuprofen, and oxycodone.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group will be asked to start with acetaminophen (650mg tablet by mouth every 6 hours) when they are in pain. If they still require additional analgesics, the second-line medication is ibuprofen (600mg tablet by mouth every 6 hours). Oxycodone (5mg tablet by mouth every 4 hours) will be the third-line medication to be used if acetaminophen and ibuprofen do not sufficiently control the pain.
  Interventions: Drug: OxyCODONE 5 Mg (milligram) Oral Tablet; Drug: Ibuprofen 600 Mg (milligram) Oral Tablet; Drug: Acetaminophen 650 MG (milligram) Oral Tablet
- Control group (Active Comparator): Patients in the control group will be asked to start with acetaminophen (650mg tablet by mouth every 6 hours) when they are in pain. If they still require additional analgesics, the second-line medication is oxycodone (5mg tablet by mouth every 4 hours).
  Interventions: Drug: OxyCODONE 5 Mg (milligram) Oral Tablet; Drug: Acetaminophen 650 MG (milligram) Oral Tablet

INTERVENTIONS:
Drug: OxyCODONE 5 Mg (milligram) Oral Tablet — Oxycodone will be the second-line treatment in the control group and the third-line treatment in the experimental group.
Drug: Ibuprofen 600 Mg (milligram) Oral Tablet — Patients in the experimental group will receive ibuprofen 600mg as the second-line analgesic.
  Arms: Experimental group
Drug: Acetaminophen 650 MG (milligram) Oral Tablet — All patients will receive acetaminophen as the first-line analgesic.

SUMMARY:
Given the ongoing national opioid epidemic, an increased interest has developed in optimizing opioid prescribing practices of physicians, including otolaryngologists. Endoscopic sinus surgery (ESS) is one of the most commonly performed surgeries by otolaryngologists with over 250,000 ESS's performed annually in the U.S. Multiple studies have shown that, compared to the amount patients actually consume, otolaryngologists prescribe a high quantity of opioids to patients recovering from ESS). It has been shown that these excess opioid medications contribute to prolonged use or abuse by the patient, family members, or friends. The purpose of this study is to better understand the pain management requirements of patients who undergo ESS for recurrent acute rhinosinusitis (RARS) or chronic rhinosinusitis (CRS).

This prospective, randomized, multi-institutional controlled trial will aim to determine the degree to which pain following ESS can be adequately controlled by non-opioid medications. It will also determine whether post-ESS narcotic use can be avoided entirely, or at least significantly limited. Patients will be randomized into two groups, each of which will receive a stepwise analgesic regimen consisting of acetaminophen and oxycodone or acetaminophen and ibuprofen. Pain will be assessed daily using visual analog scales (VAS) and the Brief Pain Inventory (BPI).

The results of this study will help to develop a standardized approach to pain management in the post-ESS setting and help to elucidate the role of non-opioid pain medications. The ultimate goal would be to positively affect opioid prescribing patterns among surgeons who perform ESS in order to significantly reduce the quantity of opioids prescribed to patients while continuing to adequately manage patients' pain.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* Scheduled to undergo endoscopic sinus surgery for sinusitis (CRSwNP, CRSsNP, or RARS)
* Can commit to follow up for at least one postoperative visit

Exclusion Criteria:

Patients undergoing a septorhinoplasty (septoplasty permissible if patient will also undergo sinus surgery)

* Doyle splints to be used
* Alcohol or opioid use disorder
* History of chronic pain disorders
* Regular use of acetaminophen/NSAIDS (>4x per week)
* Patients who use narcotics or neuromodulating drugs (e.g. gabapentin, nortriptyline)more than 2x per week on average.
* Gastrointestinal ulcers or bleeding
* Chronic kidney disease/known decreased renal function (estimated glomerular filtration rate <60)
* Liver cirrhosis or other hepatic impairment
* Prior adverse reaction to opioids or NSAIDS
* Other contraindications to any drug classes in either group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Stanford Health Care, Stanford, California
  - NorthShore University Health System, Evanston, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Albert Einstein, The Bronx, New York
  - Vanderbilt, Nashville, Tennessee
- University of British Columbia, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharyya N. Ambulatory sinus and nasal surgery in the United States: demographics and perioperative outcomes. Laryngoscope. 2010 Mar;120(3):635-8. doi: 10.1002/lary.20777. PMID 20058315
- [Background] Schwartz MA, Naples JG, Kuo CL, Falcone TE. Opioid Prescribing Patterns among Otolaryngologists. Otolaryngol Head Neck Surg. 2018 May;158(5):854-859. doi: 10.1177/0194599818757959. Epub 2018 Feb 20. PMID 29460670
- [Background] Svider PF, Arianpour K, Guo E, Folbe E, Zuliani G, Lin H, Eloy JA, Folbe AJ. Opioid prescribing patterns among otolaryngologists: Crucial insights among the medicare population. Laryngoscope. 2018 Jul;128(7):1576-1581. doi: 10.1002/lary.27101. Epub 2018 Feb 15. PMID 29446449
- [Background] Mohan S, Bhattacharyya N. Opioids and the Otolaryngologist: An Ambulatory Assessment. Otolaryngol Head Neck Surg. 2018 Jul;159(1):29-34. doi: 10.1177/0194599818765125. Epub 2018 Mar 20. PMID 29557264
- [Derived] Ayoub NF, Choby G, Turner JH, Abuzeid WM, Raviv JR, Thamboo A, Ma Y, Chandra RK, Chowdhury NI, Stokken JK, O'Brien EK, Shah S, Akbar N, Roozdar P, Nayak JV, Patel ZM, Hwang PH. Assessment of Opioid Use and Analgesic Requirements After Endoscopic Sinus Surgery: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Sep 1;147(9):811-819. doi: 10.1001/jamaoto.2021.1839. PMID 34351376

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: 1. st line analgesic: acetaminophen 650mg tablet by mouth every 6 hours
  2. nd line analgesic: ibuprofen 600mg tablet by mouth every 6 hours if they still require additional analgesics
  3. rd line analgesic: oxycodone 5mg tablet by mouth every 4 hours if they still require additional analgesics
- Control Group: 1. st line analgesic: acetaminophen 650mg tablet by mouth every 6 hours
  2. nd line analgesic: oxycodone 5mg tablet by mouth every 4 hours if they still require additional analgesics
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 56 | 62
Completed | 49 | 51
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 6 | 8
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (16.1) | 43.3 (15.9) | 46.7 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 27 | 29 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 40 | 43 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Prior sinus surgery [Count of Participants; unit: Participants] | 21 | 18 | 39
Lund-mackay score [Mean (Standard Deviation); unit: units on a scale] — The Lund-Mackay scoring system is a validated categorical scale used to define the extent of sinonasal disease on CT. The bilateral maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal sinuses are scored from 0-2, with 0 correlating to a normal sinus, 1 to partial opacification, and 2 to a fully opacified sinus. The bilateral ostiomeatal complexes are scored 0 if patent or 2 if obstructed. The total score ranges from 0 to 24, with 24 representing the most extensive disease.
  Lund VJ, Kennedy DW. Staging for rhinosinusitis. Otolaryngol Head Neck Surg 1997; 117:S35-40.
  units on a scale | 9.7 (4.8) | 11.4 (5.9) | 10.5 (5.4)
Total baseline SNOT-22 score [Mean (Standard Deviation); unit: units on a scale] — The SNOT-22 is a validated, disease-specific questionnaire in which patients report the presence and severity of 22 commonly experienced symptoms and social consequences of chronic rhinosinusitis over the prior 2-week period. Each question scales from 0 to 5, with 0 indicating "no problem" and 5 "problem as bad as it can be." The highest possible score is 110, corresponding to the most severe symptoms.
  Hopkins C, Gillett S, Black R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol 2009; 34:447-54.
  units on a scale | 39.6 (20.1) | 41.4 (19.8) | 40.5 (19.9)

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity
Description: A 10-cm visual analog scale (VAS) will be used to assess pain severity.The VAS is a continuous, patient-reported outcome measure determined using a horizontal 100-mm scale ranging from "no pain" with a score of 0 to "worst imaginable pain," corresponding to a score of 100.
Time Frame: Average pain score will be collected for preoperative visit (the day before surgery)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 12.4 (20.0) | 8.5 (13.5)

2. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Average pain score was collected for postoperative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 30.2 (26.6) | 29.4 (26.0)

3. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Average pain score will be collected for postoperative day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 27.0 (24.8) | 23.5 (23.2)

4. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Average pain score will be collected for postoperative day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 19.2 (22.6) | 22.5 (19.0)

5. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Average pain score will be collected for postoperative day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 14.1 (18.7) | 16.8 (18.1)

6. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Average pain score will be collected for postoperative day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 15.8 (21.8) | 15.0 (19.6)

7. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Average pain score will be collected for postoperative day 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 13.9 (19.0) | 11.7 (14.5)

8. Primary Outcome: Pain Severity
Description: as for outcome 1
Time Frame: Average pain score will be collected for postoperative day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 8.1 (9.8) | 10.1 (11.2)

9. Primary Outcome: Medication Log
Description: Patients kept a daily medication log and reported the number of doses consumed per day (650mg acetaminophen, 600mg ibuprofen, 5mg oxycodone). The mean number of medication doses per day was calculated for each treatment group.
Time Frame: Postoperative day 1 to 7
Measure: Mean (Standard Deviation); unit: Average number of medication doses/day
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
Average number of medication doses/day
  Oxycodone POD1 | 0.3 (0.7) | 0.6 (1.1)
  Oxycodone POD2 | 0.1 (0.3) | 0.4 (1.0)
  Oxycodone POD3 | 0.1 (0.2) | 0.3 (0.8)
  Oxycodone POD4 | 0.1 (0.3) | 0.3 (0.7)
  Oxycodone POD5 | 0.1 (0.4) | 0.3 (1.1)
  Oxycodone POD6 | 0.1 (0.3) | 0.1 (0.6)
  Oxycodone POD7 | 0 (0.2) | 0 (0.2)
  Acetaminophen POD1 | 2.0 (1.5) | 2.1 (1.8)
  Acetaminophen POD2 | 1.8 (1.4) | 1.9 (1.9)
  Acetaminophen POD3 | 1.3 (1.3) | 1.6 (1.6)
  Acetaminophen POD4 | 1.0 (1.5) | 1.5 (1.4)
  Acetaminophen POD5 | 0.9 (1.2) | 1.3 (1.4)
  Acetaminophen POD6 | 0.9 (1.3) | 1.1 (1.3)
  Acetaminophen POD7 | 0.6 (1.0) | 0.6 (0.8)
  Ibuprofen POD1 | 0.6 (0.9) | 0 (0)
  Ibuprofen POD2 | 0.5 (0.8) | 0 (0)
  Ibuprofen POD3 | 0.4 (0.9) | 0 (0)
  Ibuprofen POD4 | 0.3 (0.8) | 0 (0)
  Ibuprofen POD5 | 0.4 (0.8) | 0 (0)
  Ibuprofen POD6 | 0.3 (0.6) | 0 (0)
  Ibuprofen POD7 | 0.2 (0.5) | 0 (0)

10. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: The Brief Pain Inventory (BPI) Severity short form is a validated, patient-reported outcome measure that assesses pain over a 24-hour period. The Pain Severity score is calculated as a composite mean score using the degree of pain a patient experiences per day at its "least," "worst," "average," and "now." The score ranges from 0 to 10 (higher indicates more pain).
  Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain 2004. 20(5): 309-318.
Time Frame: BPI score will be collected at the preoperative visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 1.6 (2.2) | 1.0 (1.5)

11. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: as for outcome 10
Time Frame: Average BPI score will be collected for postoperative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 2.8 (2.3) | 2.9 (2.0)

12. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: as for outcome 10
Time Frame: Average BPI score will be collected for postoperative day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 2.5 (2.1) | 2.3 (2.0)

13. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: as for outcome 10
Time Frame: Average BPI score will be collected for postoperative day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 1.9 (2.0) | 2.1 (1.8)

14. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: as for outcome 10
Time Frame: Average BPI score will be collected for postoperative day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 1.5 (1.8) | 1.9 (1.6)

15. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: as for outcome 10
Time Frame: Average BPI score will be collected for postoperative day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 1.7 (2.1) | 1.6 (1.6)

16. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: as for outcome 10
Time Frame: Average BPI score will be collected for postoperative day 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 1.5 (1.9) | 1.4 (1.5)

17. Secondary Outcome: Brief Pain Inventory (BPI) Score
Description: as for outcome 10
Time Frame: Average BPI score will be collected for postoperative day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 1.3 (1.7) | 1.4 (1.5)

18. Secondary Outcome: Severity of Epistaxis
Description: A 10-cm visual analog scale (VAS) will be used to assess bleeding. The VAS is a continuous, patient-reported outcome measure determined using a horizontal 100-mm scale ranging from "no bleeding" with a score of 0 to "continuous bleeding," corresponding to a score of 100.
Time Frame: Epistaxis severity will be collected at the preoperative visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 0 (0) | 0 (0)

19. Secondary Outcome: Severity of Epistaxis
Description: as for outcome 18
Time Frame: Epistaxis severity will be collected for postoperative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 36.3 (33.2) | 38.9 (31.9)

20. Secondary Outcome: Severity of Epistaxis
Description: as for outcome 18
Time Frame: Epistaxis severity will be collected for postoperative day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 23.0 (27.1) | 21.6 (24.0)

21. Secondary Outcome: Severity of Epistaxis
Description: as for outcome 18
Time Frame: Epistaxis severity will be collected for postoperative day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 15.9 (22.0) | 12.9 (17.5)

22. Secondary Outcome: Severity of Epistaxis
Description: as for outcome 18
Time Frame: Epistaxis severity will be collected for postoperative day 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 9.3 (15.2) | 11.8 (16.5)

23. Secondary Outcome: Severity of Epistaxis
Description: as for outcome 18
Time Frame: Epistaxis severity will be collected for postoperative day 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 10.1 (20.1) | 7.8 (17.5)

24. Secondary Outcome: Severity of Epistaxis
Description: as for outcome 18
Time Frame: Epistaxis severity will be collected for postoperative day 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 6.5 (11.6) | 6.6 (14.1)

25. Secondary Outcome: Severity of Epistaxis
Description: as for outcome 18
Time Frame: Epistaxis severity will be collected for postoperative day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 49 | 51
units on a scale | 4.6 (9.2) | 5.4 (12.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the one week period after surgery for each participant.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

LIMITATIONS AND CAVEATS:
The low levels of narcotic consumption observed may have precluded achieving significance in pain score comparisons across groups, as the pre-hoc power analysis predicted higher levels of opioid use

Selection bias: 1) patient willingness to participate in an opioid-related study could serve as a source of bias 2) loss to follow up

Lack of blinding and placebo were additional limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT03783702/Prot_SAP_000.pdf